CLINICAL TRIAL: NCT02698293
Title: A Phase I Study of Photodynamic Therapy (PDT) Plus Vitamin D3 for High-grade Anal Dysplasia and Microinvasive Anal Cancer
Brief Title: PDT Plus Vitamin D3 for Anal Dysplasia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Covid-19
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08216
Record Dates: First submitted 2016-03-01; First posted 2016-03-03 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Anal Dysplasia; Carcinoma in Situ
MeSH Terms: conditions — Carcinoma in Situ | interventions — Cholecalciferol; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): 5-aminolevulinic acid hydrochloride (Gliolan), orally, 40 mg/kg administered approximately 4-6 hours before light administration. There will be two levels of light dose: 50 and 100 J/cm2. Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT.
  Total duration of drug product administration (including any open-label lead-in, if applicable).
  Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT.
  None This is a phase I dose escalation study, with two levels of light dose. The design is cohorts of 3s. Light at 50 Joules and Light at 100 joules There are pre-defined DLTs.
  Interventions: Drug: Gliolan; Drug: Vitamin D3 cholecalciferol); Other: Photodynamic Therpay
- Cohort 2 (Experimental): 5-aminolevulinic acid hydrochloride (Gliolan), orally, 40 mg/kg administered approximately 4-6 hours before light administration. There will be two levels of light dose: 50 and 100 J/cm2. Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT Total duration of drug product administration (including any open-label lead-in, if applicable).
  Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT.
  None This is a phase I dose escalation study, with two levels of light dose. The design is cohorts of 3s. Light at 50 Joules and Light at 100 joules There are pre-defined DLTs.
  Interventions: Drug: Gliolan; Drug: Vitamin D3 cholecalciferol); Other: Photodynamic Therpay
- Cohort 3 (Experimental): 5-aminolevulinic acid hydrochloride (Gliolan), orally, 40 mg/kg administered approximately 4-6 hours before light administration. There will be two levels of light dose: 50 and 100 J/cm2. Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT Total duration of drug product administration (including any open-label lead-in, if applicable).
  Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT.
  None This is a phase I dose escalation study, with two levels of light dose. The design is cohorts of 3s. Light at 50 Joules and Light at 100 joules There are pre-defined DLTs.
  Interventions: Drug: Gliolan; Drug: Vitamin D3 cholecalciferol); Other: Photodynamic Therpay

INTERVENTIONS:
Drug: Gliolan — orally, 40 mg/kg 4-6 hours prior to light application
  Other Names: ALA
Drug: Vitamin D3 cholecalciferol) — Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT.
  Other Names: Natures Made Vitamin D3
Other: Photodynamic Therpay — Approximately 4-6 hours after photosensitizer administration, activating light will be applied.
  The target mucosal lesion will be identified based on the initial clinical evaluation. Treatment light will be generated using a Modulight ML7710-630-6K diode laser, This laser produces up to 6W total power, with a peak wavelength of 630nm and 90% of laser power within 630-633 nm.
  The light fluence (doses) will be 50 and 100 Joules per square centimeter.
  Other Names: PDT

SUMMARY:
This is a phase I dose escalation study of photodynamic therapy (PDT) for the treatment of patients with pre-malignant tumors and superficial microinvasive disease of the anal canal and/or perianal skin. All subjects (a maximum of 12) will be given the photosensitizer ALA orally followed by the administration of red light (629-635 nm) to the tumor from a laser. The dose of ALA will be 40 mg/kg administered approximately 4-6 hours before light administration. There will be two levels of light dose: 50 and 100 J/cm2, 3-6 patients in each. Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT. Patients will be observed for 30 days for the development of DLT. Patients will be followed up for 24 months for additional toxicity and efficacy data collection.

DETAILED DESCRIPTION:
This is a phase I dose escalation study of photodynamic therapy (PDT) for the treatment of patients with pre-malignant tumors and superficial microinvasive disease of the anal canal and/or perianal skin. All subjects (a maximum of 12) will be given the photosensitizer ALA orally followed by the administration of red light (629-635 nm) to the tumor from a laser. The dose of ALA will be 40 mg/kg administered approximately 4-6 hours before light administration. There will be two levels of light dose: 50 and 100 J/cm2, 3-6 patients in each. Vitamin D3 (cholecalciferol) supplementation (10,000 IU daily) will be provided from 3 days prior through 14 weeks after light delivery for PDT. Patients will be observed for 30 days for the development of DLT. Patients will be followed up for 24 months for additional toxicity and efficacy data collection.

ELIGIBILITY:
Inclusion Criteria

* A histological or cytological diagnosis of high-grade dysplasia or carcinoma in-situ, within past 4 months.
* Premalignant lesions containing focal microinvasion are eligible when:

  * Surgery is not clinically mandated.
  * Subjects with medical conditions precluding surgery.
  * Subjects whose lesions cannot be completely resected based on size or location, or where significant functional morbidity would be anticipated with further surgery.
  * Patients refuse surgery.
* The justification for inclusion of patients with microinvasive disease is based reports demonstrating the ability of photodynamic therapy to successfully treat both dysplasia and T1 squamous cell carcinoma of the anal canal
* HPV positive by Cobas or other cytological assays within past 4 months
* Documented HIV positivity
* Patients must be on highly active anti-retroviral therapy with a CD4 count >200 for the past 12 months
* Viral load <200 for 12 months for the past 12 months
* ECOG performance status of 0-1.
* 18 years of age or older.
* Study subjects capable of providing informed consent.
* Women of childbearing potential and men must agree to use a medically accepted method of birth control from the time they sign consent and until one month after receiving ALA

Exclusion Criteria:

* Study subjects in whom the lesion has invasive squamous cell carcinoma of the anal cavity which is clinically appreciable.
* Clinically occult microinvasive squamous cell carcinoma of the anal cavity which is not focal.
* Study subjects who are pregnant or lactating .
* Study subjects who have a platelet count of less than 100,000/cubic mm.
* Study subjects with elevated aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, or total bilirubin levels >2X normal or a history of chronic liver disease or cirrhosis of the liver.
* Significant cardiovascular history that would put the study subject at risk from hypotension that may occur with ALA
* Study subjects with porphyria or hypersensitivity to porphyrins.
* Administration of the following compounds: tetracyclines, sulfonamides, fluoroquinolones within 48 hours, or hypericin extracts within a week prior to light administration.
* Study subjects with abnormal baseline creatinine level or diagnosed kidney disease.
* Treatment with 5-FU, Imiquimod, trichloroacetic acid or ablative therapy within the previous month.
* Study subjects who have a medical history of immune suppression. This will include patients with a past transplantation requiring ongoing immunosuppressive medications.
* A history of sarcoidosis, hyperphosphatemia, or known kidney stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | 18 months
  DLTs have been defined

CONTACTS AND LOCATIONS:
Overall Officials: Keith Cengel, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No